CLINICAL TRIAL: NCT06554795
Title: A Phase 1/2a, Multicenter, Open-Label, First in Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of DB-1419 in Participants With Advanced/Metastatic Solid Tumors
Brief Title: First-in-human Study of DB-1419 for Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DB-1419-O-1001
Record Dates: First submitted 2024-08-06; First posted 2024-08-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Dose Level 1 (Experimental): Enrolled subjects will receive DB-1419 at Dose Level 1
  Interventions: Drug: DB-1419
- Dose Level 2 (Experimental): Enrolled subjects will receive DB-1419 at Dose Level 2
  Interventions: Drug: DB-1419
- Dose Level 3 (Experimental): Enrolled subjects will receive DB-1419 at Dose Level 3
  Interventions: Drug: DB-1419
- Dose Level 4 (Experimental): Enrolled subjects will receive DB-1419 at Dose Level 4
  Interventions: Drug: DB-1419
- Dose Level 5 (Experimental): Enrolled subjects will receive DB-1419 at Dose Level 5
  Interventions: Drug: DB-1419
- Dose Level 6 (Experimental): Enrolled subjects will receive DB-1419 at Dose Level 6
  Interventions: Drug: DB-1419
- Dose Expansion 1 (Experimental)
  Interventions: Drug: DB-1419
- Dose Expansion 2 (Experimental)
  Interventions: Drug: DB-1419
- Dose Expansion 3 (Experimental)
  Interventions: Drug: DB-1419
- Dose Expansion 4 (Experimental)
  Interventions: Drug: DB-1419
- Dose Expansion 5 (Experimental)
  Interventions: Drug: DB-1419
- Dose Expansion 6 (Experimental)
  Interventions: Drug: DB-1419
- Dose Expansion 7 (Experimental)
  Interventions: Drug: DB-1419
- Dose Expansion 8 (Experimental)
  Interventions: Drug: DB-1419

INTERVENTIONS:
Drug: DB-1419 — Administered Injection of Vein (I.V.)

SUMMARY:
A Phase 1/2a First-in-Human Study of DB-1419 in Advanced/Metastatic Solid Tumors

DETAILED DESCRIPTION:
A Phase 1/2a, Multicenter, Open-Label, First in Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of DB-1419 in Participants with Advanced/Metastatic Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 years at the time of voluntarily signing informed consent.
2. Histologically or cytologically confirmed unresectable advanced/metastatic solid tumor that has relapsed or progressed on or after standard systemic treatments, or refused the standard treatment, or for which no standard treatment is available.
3. At least one measurable lesion as assessed by the Investigator according to RECIST v1.1 criteria (Only applicable to backfill participants in phase 1a and participants in phase 1b/2a). CRPC participants with bone-only disease may be eligible on a case-by-case basis after discussion with the Medical Monitor.
4. Has a life expectancy of ≥ 3 months.
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
6. Has LVEF ≥ 50% by either echocardiography (ECHO) or multiple-gated acquisition (MUGA) within 28 days before enrollment.
7. Has adequate organ function within 7 days prior to the first dose of study treatment.
8. Has adequate treatment washout period prior to the first dose of study treatment.
9. Is willing to provide pre-existing resected tumor samples when available or undergo fresh tumor biopsy if feasible for the measurement of B7-H3/PD-L1 level and other biomarkers if no contraindication.

   Note: there is no minimum B7-H3/PD-L1 expression level mandatory for entry into the study.
10. Is capable of comprehending study procedures and risks outlined in the informed consent and able to provide written consent and agree to comply with the requirements of the study and the schedule of assessments.

Exclusion Criteria:

1. Prior treatment with B7-H3 targeted therapy.
2. Has a medical history of symptomatic congestive heart failure (New York Heart Association [NYHA] classes II-IV or serious cardiac arrhythmia requiring treatment.
3. Has a medical history of myocardial infarction or unstable angina within 6 months before enrollment.
4. Has an average of Fredericia's formula-QT corrected interval (QTcF) prolongation to > 470 millisecond (ms) in males and females based on a 12-lead electrocardiogram (ECG) in triplicate.
5. Has a medical history of interstitial lung diseases (e.g., non-infectious interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis which needs glucocorticoids and antibiotics) or current interstitial lung diseases or who are suspected to have these diseases by imaging at screening.
6. Has a history of underlying pulmonary disorder including, but not limited to, pulmonary emboli within 3 months of the start of study treatment, severe asthma, severe COPD, restrictive lung disease, and other clinically significant pulmonary compromise or requirement for supplemental oxygen.
7. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed.
8. Has an uncontrolled infection requiring intravenous injection of antibiotics, antivirals, or antifungals within 2 weeks before first dose of study treatment.
9. Know human immunodeficiency virus (HIV) infection.
10. Has spinal cord compression or clinically active central nervous system (CNS) metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Participants with asymptomatic CNS metastases who are radiologically and neurologically stable for at least 4 weeks following CNS-directed therapy (defined as 2 brain images, same imaging modality, both of which are obtained after treatment to the brain metastases; these imaging scans should be obtained at least 4 weeks apart and show no evidence of intracranial progression), and are on stable or decreasing doses of corticosteroids equivalent to ≤10 mg/day prednisone are eligible for study entry.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1/2a: Percentage of Participants with Adverse events (AE) serious AE (SAE) | Up to 30 days after last study treatment administration or before starting new anticancer treatment, whichever comes first
  Percentage of participants with TEAEs graded according to NCI CTCAE v5.0
Phase 1/2a: Percentage of Participants with serious AE (SAE) | Up to 30 days after last study treatment administration or before starting new anticancer treatment, whichever comes first
  Percentage of participants with SAEs graded according to NCI CTCAE v5.0
Phase 1a: Maximum Tolerated Dose (MTD) | From first study treatment administration until the initiation of Phase1b/2a, approximately up to 12 months.
  MTD on the data collected during Part 1
Phase 1a: Recommended Phase 2 Dose (RP2D) | From first study treatment administration until the initiation of Phase 1b/2a, approximately up to 12 months.
  RP2D of DB-1419 based on the data collected during Part 1
Phase 1b/2a: Objective Response Rate (ORR) determined by Investigator per RECIST v1.1 | Up to disease progression or death or before starting new anticancer treatment or withdrawal from the trial, whichever comes first, approximately up to 12 months.
  The percentage of subjects who had a best response rating of CR and PR

SECONDARY OUTCOMES:
Phase 1a: ORR determined from tumor assessments by Investigator per RECIST v1.1 | Up to disease progression or death or before starting new anticancer treatment or withdrawal from the trial, whichever comes first, approximately up to 12 months.
  The percentage of subjects who had a best response rating of CR and PR
Phase 1/2a: Progression free survival (PFS) determined from tumor assessments by Investigator per response evaluation criteria in solid tumors version 1.1 (RECIST v1.1 | Up to disease progression or death or before starting new anticancer treatment or withdrawal from the trial, whichever comes first, approximately up to 12 months
  PFS will be determined from tumor assessments by investigator per RECIST 1.1
Phase 1/2a: OS | From the start date of study drug to the date of death due to any cause, whichever occurs first, approximately up to 12 months after last patient first dose.
  overall survival (OS)
Phase 1/2a: AUC0-last | within 8 cycles (each cycle is 21 days or 14 days)
  the area under the concentration-time curve from time zero to the last quantifiable concentration
Phase 1/2a: AUC0-tau | within 8 cycles (each cycle is 21 days or 14 days)
  the area under the concentration-time curve from time zero to time tau
Phase 1/2a: AUCinf | within 8 cycles (each cycle is 21 days or 14 days)
  the area under the concentration-time curve from time zero to infinite
Phase 1/2a: Cmax | within 8 cycles (each cycle is 21 days or 14 days)
  peak observed concentration
Phase 1/2a: Tmax | within 8 cycles (each cycle is 21 days or 14 days)
  Time to Cmax
Phase 1/2a: Ctrough | within 8 cycles (each cycle is 21 days or 14 days)
  trough concentration
Phase 1/2a: ADA prevalence | within 8 cycles (each cycle is 21 days or 14 days)
  the proportion of participants who are ADA positive at any point in time (at baseline and post-baseline)
Phase 1/2a: ADA incidence | within 8 cycles (each cycle is 21 days or 14 days)
  the proportion of participants having treatment-emergent ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hu, Study Director — DualityBio Inc.
Locations (33):
- United States (10):
  - Site USA12-0, Los Angeles, California
  - Site USA08-0, Newport Beach, California
  - Site USA13-0, Sacramento, California
  - Site USA06-0, Washington D.C., District of Columbia
  - Site USA02-0, Florida City, Florida
  - Site USA11-0, Chicago, Illinois
  - Site USA03, Huntersville, North Carolina
  - Site USA05-0, Philadelphia, Pennsylvania
  - Site USA07-0, Nashville, Tennessee
  - Site USA09-0, West Valley City, Utah
- Australia (3):
  - AUS03-0, North Ryde, New South Wales
  - AUS01-0, Randwick, New South Wales
  - AUS02-0, Nedlands, Western Australia
- China (20):
  - Site CHN24-0, Hefei, Anhui
  - Site CHN28-0, Beijing, Beijing Municipality
  - Site CHN16-0, Chongqing, Chongqing Municipality
  - Site CHN20-0, Fuzhou, Fujian
  - Site CHN32-0, Nanning, Guangxi
  - Site CHN08-0, Harbin, Heilongjiang
  - Site CHN23-0, Harbin, Heilongjiang
  - Site CHN03-0, Luoyang, Henan
  - Site CHN09-0, Zhengzhou, Henan
  - Site CHN25-0, Zhengzhou, Henan
  - Site CHN21-0, Changsha, Hunan
  - Site CHN29-0, Jinan, Shandong
  - Site CHN26-0, Linyi, Shandong
  - Site CHN01-0, Shanghai, Shanghai Municipality
  - Site CHN15-0, Shanghai, Shanghai Municipality
  - Site CHN18-0, Chengdu, Sichuan
  - Site CHN38-0, Tianjin, Tianjin Municipality
  - Site CHN19-0, Kunming, Yunnan
  - Site CHN17-0, Hangzhou, Zhejiang
  - Site CHN37-0, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li C, Yao J, Yang J, Zhang Y, Qiu Y, Zhu Z, Hua H. Preclinical Evaluation of DB-1419, a Novel Bifunctional and Bispecific Anti-B7-H3 x PD-L1 Antibody-Drug Conjugate. Clin Cancer Res. 2025 Aug 14;31(16):3581-3593. doi: 10.1158/1078-0432.CCR-25-0634. PMID 40499141